CLINICAL TRIAL: NCT06887881
Title: Clinical Use of Preimplantation DNA Methylation Screening (PIMS) and Preimplantation Genetics Screening (PGT-A) in Infertile PCOS Patients-A Multicenter, Prospective Randomized Non-inferior Clinical Trial
Brief Title: PIMS vs PGT-A in Infertile PCOS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: The Third Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Provincial Maternal and Child Health Hospital (Other); Guangzhou Medical University Affiliated Women and Children's Medical Center (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University Shenzhen Hospital (Other); BoAi Hospital of Zhongshan (Other); Zhuhai Maternal and Child Health Hospital (Unknown); Shenzhen Maternal and Child Health Hospital (Unknown); Liuzhou Hospital of Guangzhou Women and Children's Medical Center (Unknown); Guangxi Zhuang Autonomous Region Maternal and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Zhou Canquan, Chief Physician, professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: [2024]345-2
Record Dates: First submitted 2024-01-25; First posted 2025-03-20 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: PGT-A; PCOS; PIMS
Keywords: PIMS; PCOS; PGT-A; cumulative live birth rate; early pregnancy loss rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMS Group (Experimental): Couples in the PIMS group will have up to 6 blastocysts screened with PIMS and a single euploid embryo with the optimal state of whole-genome DNA methylation and the highest morphologic score will be selected for the initial transfer. The optimal state of whole-genome DNA methylation includes methylation level closest to the optimal level (0.26 according to our preliminary results) and proper methylation state for some specific regions.Blastocysts that have undergone a second biopsy will not be preferred.
  Interventions: Genetic: PIMS screening
- PGT-A Group (Active Comparator): Couples in the PGT-A group will have up to 6 blastocysts screened with PGT-A and a single euploid blastocyst with the highest morphologic score selected for the initial transfer.Blastocysts that have undergone a second biopsy will not be preferred.
  Interventions: Genetic: PGT-A screening

INTERVENTIONS:
Genetic: PIMS screening — Couples in the PIMS group will have up to 6 blastocysts screened with PIMS and a single euploid embryo with the optimal state of whole-genome DNA methylation and the highest morphologic score will be selected for the initial transfer
  Arms: PIMS Group
Genetic: PGT-A screening — Couples in the PGT-A group will have up to 6 blastocysts screened with PGT-A and a single euploid blastocyst with the highest morphologic score selected for the initial transfer.
  Arms: PGT-A Group

SUMMARY:
This experiment has become a serious issue for two reasons: DNA methylation plays an important role during embryogenesis, global abnormal methylome reprogramming often occurs in human embryos, and DNA methylome pattern is associated with live birth rate. The endocrine metabolic disorders of polycystic ovarian syndrome (PCOS) patients may affect the epigenetic status of embryos and lead to the increase of early pregnancy loss rate in PCOS patients. However, there is still no technology using DNA methylome as an indicator in preimplantation embryo screening in PCOS patients. Our recent study showed that using Pre-implantation Methylation Screening (PIMS) can select embryos with better methylation state and euploid chromosomes. The efficiency of PIMS in PCOS patients needs further validation through randomized controlled clinical trial.

The purpose of the study is to compare whether the two groups of PCOS patients who selected embryos using PIMS and selected embryos using "PGT-A + morphology"had any difference in early pregnancy loss rate. This study aims to explore whether PIMS can be used as another embryo evaluation method besides "PGT-A+morphology" to screen good developmental potential embryos in patients with PCOS. Investigators need to clarify whether a better embryo evaluation system can be established through PIMS technology during assisted reproductive treatment for infertile PCOS couples and provide credible and effective evidence-based medical evidence for the application of PMIS technology in the field of reproductive medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 20 and 40 years diagnosed with PCOS according to international evidence-based guidline for assessment and management of policystic ovarian syndrome 2018.
2. Women who plan to undergo the 1st/2nd IVF/ICSI/PGT-A treatment cycle.
3. Women who obtain 2 or more blastocysts that have morphological score of 4BC/4CB or better on Day 5of embryo culture.
4. Culture all the cleavage stage embryos into blastocysts, conduct biopsy on all the blastocysts, and cryopreserve each blastocyst as a single embryo
5. Agree to the thawing and transfer of a single blastocyst.
6. Sign the informed consent form.

Exclusion Criteria:

1. Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus unicornate, bicornate, or duplex); untreated uterine septum, submucous myoma, or endometrial polyp(s); or with history of intrauterine adhesions.
2. Women who are indicated and planned to undergo preimplantation genetic testing for structural rearrangements (PGT-SR) or preimplantation genetic testing for monogenic (PGT-M).
3. Women who use donated oocytes or sperm to achieve pregnancy.
4. Women with contraindication for assisted reproductive technology or for pregnancy, such as undiagnosed liver disease or dysfunction (based on serum liver enzyme testing); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; uncontrolled hypertension, known symptomatic heart disease; history of or suspected carcinoma including including cervical carcinoma, endometrial carcinoma, or breast carcinoma; undiagnosed vaginal bleeding and so on.
5. Untreated hydrosalpinx according to ultrasonography test.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 766 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
early pregnancy loss rate | From enrollment to the end of treatment at 12months
  early pregnancy loss rate in one year after randomization
cumulative live birth rate per oocyte retrieval cycle | From enrollment to the end of treatment at 12months
  cumulative live birth rate per oocyte retrieval cycle in one year after randomization

SECONDARY OUTCOMES:
clinical pregnancy rate after initial embryo transfer | From enrollment to the end of treatment at 12months
time to get live birth | From enrollment to the end of treatment at 12months
the rate of a Good Birth Outcome | From enrollment to the end of treatment at 12months
multiple pregnancy rate | From enrollment to the end of treatment at 12months
duration of pregnancy | From enrollment to the end of treatment at 12months
birth weight | From enrollment to the end of treatment at 12months
incidence of maternal and neonatal complications (including fetal anomalies) | From enrollment to the end of treatment at 12months